CLINICAL TRIAL: NCT07171658
Title: Improving Cervical Cancer Screening Coverage Among Underscreened Women Aged 50 to 74 in Switzerland Using HPV Self-sampling Strategies: A Randomized Study - Breast Cancer-Related Approach for Increasing Cervical Cancer Screening
Brief Title: Breast Cancer-Related Approach for Increasing Cervical Cancer Screening
Acronym: BRAICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Di Vincenzo Sormani (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Jessica Di Vincenzo Sormani, Professor assistant (tenure track), School of Health Sciences Geneva
Organization: School of Health Sciences Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 32HW-0_228666
Record Dates: First submitted 2025-08-25; First posted 2025-09-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer Screening
Keywords: cervical cancer screening; underscreened women; HPV self-sampling; Integrated approach
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: The study is a 1) population-based 2) randomized trial 3) two-arm 4) open 5) national hybrid 6) completed by an observational control arm .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group 1: Sensitization to Cervical Cancer (CC) screening (Experimental): Women will receive an awareness letter explaining the importance of cervical cancer screening, the Swiss recommendations and an invitation to schedule an appointment.
  Interventions: Behavioral: Sensitization to Cervical Cancer (CC) screening
- Intervention Group 2: Home-based HPV self-sampling (Experimental): Women will receive a free-of-charge vaginal self-sampling kit for HPV infection.
  Interventions: Behavioral: Home-based HPV self-sampling

INTERVENTIONS:
Behavioral: Sensitization to Cervical Cancer (CC) screening — Women will receive an awareness letter explaining the importance of cervical cancer screening, the Swiss recommendations and an invitation to schedule an appointment.
  Arms: Intervention Group 1: Sensitization to Cervical Cancer (CC) screening
Behavioral: Home-based HPV self-sampling — Women will receive a free-of-charge vaginal self-sampling kit for HPV infection.
  Arms: Intervention Group 2: Home-based HPV self-sampling

SUMMARY:
The primary objective of this clinical trial is to assess cervical cancer screening participation among under-screened women invited through organized breast cancer screening programs in Switzerland.

This randomized trial will compare three arms:

1. Intervention group 1: Sensitization to Cervical Cancer (CC) screening Women will receive an awareness letter explaining the importance of cervical cancer screening, the Swiss recommendations and an invitation to schedule an appointment.
2. Intervention group 2: Home-based Human papillomavirus infection (HPV) self-sampling Women will receive a free-of-charge vaginal self-sampling kit for HPV infection
3. Observational control group Women selected in the control arm will only be recruited one year following the screening of those in the intervention arm (T0+1), as to not influence Cervical Cancer Screening (CCS) behavior during this period by being reminded of screening recommendations.

DETAILED DESCRIPTION:
Secondary objectives are:

* To identify and compare the association of socio-demographic characteristics with screening participation in all study arms (cf. 3.2 study design).
* To compare the use of primary screening methods (HPV test vs. Papanicolaou test) between study arms.
* To compare prevalence of positive primary screening and triage results between study arms.
* To compare follow-up rates for participants screened positive in both intervention arms.
* To evaluate acceptability of both screening strategies (sensitization vs. home-based).
* To assess the relationship between CCS behavior and Breast Cancer Screening (BCS) behavior.

ELIGIBILITY:
Inclusion Criteria:

* Women receiving Breast Cancer Screening (BCS) invitation letters in the selected five cantons (Geneva, Bern (francophone), Jura, Neuchâtel, and Vaud)
* Aged 50 to 74 years old
* Not been screened for cervical cancer in the past three years
* Speaking one of the 6 languages of the study (French, German, Italian, and in English, Spanish, and Portuguese)

Exclusion Criteria:

* Prior cervical cancer diagnosis,
* Hysterectomy
* Non consent to participate to the study
* Incapable of judgment or under tutelage
* Pregnancy

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation to Cervical Cancer Screening (CCS) | 12 months
  Participation to Cervical Cancer Screening (CCS) (primary HPV test or cytology) in the past 12 months, self-declared, proportion in %

SECONDARY OUTCOMES:
Correlation of socio-demographic characteristics with screening participation | 12 months
  Regression coefficients of screening in the past 12 months for: education level, occupation, relationship status, sexual orientation, mother tongue, country of origin, residential area, children, follow-up by general practitioner or gynecologist, age, number of years living in Switzerland, Body Mass Index (calculated based on weight and height).
  Measurement tool: self-reported from questionnaire
Choice of primary screening methods (HPV testing vs cytology) | 12 months
  Difference between study arms of the proportion of participants screened by HPV test versus cytology in each arm.
Prevalence of positive primary screening (HPS test) and triage results (cytology) | 12 months
  Difference between study arms of the:
  * Prevalence of screen-positive women (i.e. HPV-positive or Atypical squamous cells of undetermined significance - ASC-US+)
  * Proportion (%) of HPV-positive women with ASC-US+ upon triage
  * Proportion (%) of Cervical Intraepithelial Neoplasia Grade 2 (CIN2+) diagnosed
  * Proportion (%) of Cervical Cancer (CC) diagnosed
  * Proportion (%) of participants treated for CIN2+ or CC
Follow-up rates for participants screened positive | 12 months
  Difference between study arms of the proportion (%) of primary screen-positive women who have undergone triage
Acceptability of screening strategies | 12 months
  Difference between study arms of the:
  - Mean satisfaction score (Likert scale, from 1 Totalement satisfied to 4 Very unsatisfied)
Reasons for non-compliance | 12 months
  Proportion (%) of participants among unscreened women indicating predefined reasons for non-compliance
Association between Cervical Cancer Screening (CCS) behavior and Breast Cancer Screening (BCS) screening behaviors | 12 months
  Difference in the study arms: of the proportion (%) of participants having done all screenings, and participants having selected only one or two screenings, and participants having done none.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Di Vincenzo Sormani, PhD, Study Director — Haute École de Santé de Genève (HEdS-GE)
Locations (1):
- University Hospitals of Geneva, Geneva, Canton of Geneva, Switzerland